CLINICAL TRIAL: NCT00693758
Title: Magnetic Resonance Imaging for the Detection of Oxygen Changes in the Heart
Brief Title: Assessment of Oxygen Changes in the Heart With Cardio-vascular Magnetic Resonance Imaging
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Oliver Strohm, Adunct Research Associate Professor, University of Calgary
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18798; 18798
Record Dates: First submitted 2007-12-10; First posted 2008-06-09 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Vascular Diseases; Myocardial Ischemia
Keywords: MRI; coronary reactivity; coronary physiology
MeSH Terms: conditions — Vascular Diseases; Myocardial Ischemia | interventions — Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (No Intervention): healthy volunteers without intervention
  Interventions: Device: Breathing gas
- 2 (No Intervention): patients with suspected coronary artery disease without intervention
- 3 (Experimental): Healthy volunteers during adenosine infusion
  Interventions: Drug: adenosine; Device: Blood pressure cuff
- 4 (Experimental): Healthy volunteers during changes of breathing gases (CO2, O2)
  Interventions: Other: modified end-tidal forcing system
- 5 (Experimental): patients with suspected coronary artery disease during adenosine infusion
  Interventions: Drug: adenosine
- 6 (Experimental): patients with suspected coronary artery disease during changes of breathing gases
  Interventions: Other: modified end-tidal forcing system
- 7 (Experimental): Assessment of reactive hyperemia in arms of healthy volunteers to improve sequences
  Interventions: Other: arm cuff occlusion

INTERVENTIONS:
Drug: adenosine — intravenous infusion of adenosine (140microgr./min/kg)
  Other Names: Adenosine stress
  Arms: 3; 5
Other: modified end-tidal forcing system — changes in partial pressures of O2 and CO2 in inspired air
  Other Names: O2 / CO2 changes in inspired air
  Arms: 4; 6
Other: arm cuff occlusion — 3 min. lasting upper arm cuff occlusion
  Arms: 7
Device: Breathing gas — Changes in pO2 and pCO2 in inspired air mix
  Arms: 1
Device: Blood pressure cuff — supra-systolic arm occlusion with pressure cuff
  Arms: 3

SUMMARY:
The ability of a new SSFP-based BOLD MRI sequence to assess myocardial oxygenation changes in response to coronary flow changes induced by adenosine and increased CO2-partial pressure will be examined in healthy volunteers and patients with suspected coronary artery disease. Also the susceptibility of a new SSFP-based BOLD sensitive MRI sequence to changes in arterial oxygenation will be examined. This will help understand the physiologic basis of oxygen sensitive imaging of the heart.

DETAILED DESCRIPTION:
A new SSFP based T2 and T2* sensitive sequence which provides good BOLD contrast will be used. It was developed by researchers at the Stephenson CMR Centre and Northwestern University of Chicago. Its major advantage to previous BOLD sensitive sequences is its lower susceptibility to motion artifacts.

MR imaging is performed with a commercial 1.5 T Siemens MR scanner (Siemens Avanto). In order to obtain a homogeneous magnetic field an additional surface chest coil is used in combination to the body coil. Three short axis views representing basal, mid and apical slices are set up and are used throughout the study. If the volunteer has to be moved from their position for any reason, similar short axis views will be attempted.

In order to improve and further develop the MRI sequence the technique will be used in a arm-cuff model in healthy volunteers, using reactive hyperemia, which is easier to image than the heart. The BOLD-MRI signal intensity of the forearm will be assessed during a short, 3 min. lasting upper arm-cuff occlusion and the following reactive hyperemia.

Main interest of the study is the examination of the heart of healthy volunteers as well as patients with suspected coronary heart disease with this BOLD-MRI technique. The signal intensity of the myocardium at rest and after different coronary flow stimulation will be assessed. These stimuli will be pharmacologic (adenosine) as well as changes in arterial CO2 and O2 pressure.

All subjects that will undergo changes in their breathing gases, will first be examined in the vascular research laboratory of Dr. M. Poulin. There the subjects will be familiarized with the modified end-tidal forcing system (MEFS) and their individual response to changes in breathing gases will be assessed. A complete dry-run of the breathing protocol will be performed including 2 capillary blood gas analysis. On a second day subjects will be studied in the temperature-controlled MR scanning room at Stephenson CMR Centre in a fasting state for the previous 4 hours. This includes refrain from caffeine and nicotine in these preceding 4 hours. Prior to baseline scanning, capillary blood will be sampled from the finger for blood gas, hemoglobin and hematocrit analysis. Thereafter, the volunteer will be connected to the MEFS. A baseline scan will then be performed comprising of localization, cine imaging, cross sectional flow measurement of the coronary sinus (CS) and BOLD MRI of three representative short axis slices. Then an intravenous adenosine infusion will be started. After 3 min. MR scan will be repeated. After 5 min. of rest another baseline will be recorded. Then successively the carbon dioxide pressure will be increased in two steps to 40 and 45 mmHg. After a resting period of 5 min, another baseline scan will be performed. Then oxygen partial pressure of the inspired air will be reduced in 3 steps as described in the following paragraph until an inspiratory oxygen partial pressure of 45 mmHg is achieved. This will reflect an arterial oxygen saturation of approximately 90, 85 and 80%. At each step, BOLD MRI (3 axial slices) and cross sectional flow measurements of CS will be performed. Following 5 minutes of rest another baseline scan will be performed. Throughout experimentation the subject will be connected to the METFS and we will measure ventilation, blood pressure (noninvasive), heart rate (electrocardiogram) and arterial oxygen saturation (pulse oximetry).

Image-analysis: A region of interest will be drawn around the myocardium of each short axis. The averaged signal intensity is assessed and compared to baseline after adenosine infusion and at the different levels of arterial oxygenation and carbon dioxide concentration. Additionally, differential analysis for subendocardium and subepicardium will be performed.

Coronary flow in the coronary sinus will be calculated using phase contrast MRI. This technique was first described by van Rossum, validated in phantoms and animal studies and successfully used in human patient studies. Because of the relatively small diameter of the CS, absolute flow values may not be very accurate; therefore the relative change between different levels of hypoxia will be calculated.

End-points:

BOLD SI in the myocardium defined as the averaged signal intensity of the myocardium.

Relative flow changes in CS to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent
* age > 18 years
* no known cardiovascular disease and no vasoactive medication (if recruited as healthy volunteer)
* suspected coronary artery disease or microvascular dysfunction (if recruited as patient)
* no known obstructive or restrictive lung disease
* fasting for 4 hours prior to the study

Exclusion Criteria:

* Contraindications for MRI
* Known obstructive or restrictive lung disease
* concomitant serious medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
BOLD-MRI signal intensity changes | 60

SECONDARY OUTCOMES:
Flow changes | 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Friedrich, MD, Principal Investigator — University of Calgary
Locations (1):
- Stephenson CMR Centre at Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada